CLINICAL TRIAL: NCT04140357
Title: Is There a Role for Ultrasonography in the Airway Management of Patients With Obesity
Brief Title: Role of Ultrasonography in Airway Management
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, başak gülel, Principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: BasakUltrasonografi
Record Dates: First submitted 2019-10-16; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Obese Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ultrasound is one of the most useful devices in daily anesthesia practice. Latest purpose of ultrasound usage is prediction of difficult intubation. In this study, we aimed to predict difficult laryngoscopy and intubation by using ultrasound measurement of neck soft tissue thickness in obese patient preoperatively.

DETAILED DESCRIPTION:
In this prospective and randomized controlled study, mallampati scores, interincisor gap, thyromental distance, neck circumference measurement and upper lip bite test scores will be recorded in sixty obese patients.

Additionally, neck tissue thickness will be recorded at 4 different levels (hyoid bone-skin distance, epiglot-skin distance , thyroid istmus-skin distance, vocal cord-skin distance) after the sniffing position by ultrasound with the linear probe. All measurements will be repeated three times and an average values will be recorded.

After all this measurements, endotracheal intubation will be performed by an experienced anesthetist who is uninformed about study. During intubation the Cormack Lehane (C/L, grade 1: full view of the vocal cords; grade 2a: partial view of the glottis; 2b: posterior part of the vocal cord and arytenoids visible; grade 3: only epiglottis visible; and grade 4: neither epiglottis nor glottis visible) and the Intubation Difficulty Scale (IDS) score (the numbers of attempts, operators, and alternative techniques used, the C/L grade of laryngoscopic view, lifting force and external laryngeal manipulation required, and position of the vocal cords. Every insertion of the laryngoscope and advancement of the tracheal tube towards the glottis counted as an attempt. A score of >5 indicates moderate-to-major difficulty) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30
* 18-65 YEARS
* ASA 1-2-3
* Obese patients

Exclusion Criteria:

* Pregnancy
* Upper airway pathology
* Cervical spine pathology
* Laryngeal pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with obesity body mass index >30 undergoing surgery and requiring tracheal intubation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Hyoid bone-skin distance -effect of ultrasound on prediction of difficult laryngoscopy | 30 minutes before induction
  The hyoid bone-skin distance will be measured by using ultrasound in centimeters
Epiglottis-skin distance | 30 minutes before induction
  The epiglottis-skin distance will be measured by using ultrasound in centimeters
Thyroid isthmus-skin distance | 30 minutes before induction
  The thyroid isthmus-skin distance will be measured by using ultrasound in centimeters
Vocal cord-skin distance | 30 minutes before induction
  The vocal cord-skin distance will be measured by using ultrasound in centimeters

SECONDARY OUTCOMES:
Intubation difficulty scale score | 1 minutes after intubation
  Each number of numbers attempt, operator and alternative techniques used, the Cormack Lehane score of laryngoscopic view, lifting force and external laryngeal manipulation required, and position of the vocal cords count 1 point. A score of >5 indicates moderate-to-major difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Basak Gulel, Principal Investigator — Sbü Dışkapı Yıldırım Beyazıt Eğitim Ve Araştırma Hastanesi
Locations (1):
- Başak Gülel, Ankara, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Qasmi A, Al-Alawi W, Malik AM, Manzoor Khan R, Kaul N. Comparison of Tracheal Intubation Using the Storz's C-Mac D-blade(TM) Video-Laryngoscope Aided by Truflex(TM) Articulating Stylet and the Portex(TM) Intubating Stylet. Anesth Pain Med. 2015 Dec 5;5(6):e32299. doi: 10.5812/aapm.32299. eCollection 2015 Dec. PMID 26705531
- [Result] Wu J, Dong J, Ding Y, Zheng J. Role of anterior neck soft tissue quantifications by ultrasound in predicting difficult laryngoscopy. Med Sci Monit. 2014 Nov 18;20:2343-50. doi: 10.12659/MSM.891037. PMID 25403231
- [Result] Ezri T, Gewurtz G, Sessler DI, Medalion B, Szmuk P, Hagberg C, Susmallian S. Prediction of difficult laryngoscopy in obese patients by ultrasound quantification of anterior neck soft tissue. Anaesthesia. 2003 Nov;58(11):1111-4. doi: 10.1046/j.1365-2044.2003.03412.x. PMID 14616599
- [Result] Shiga T, Wajima Z, Inoue T, Sakamoto A. Predicting difficult intubation in apparently normal patients: a meta-analysis of bedside screening test performance. Anesthesiology. 2005 Aug;103(2):429-37. doi: 10.1097/00000542-200508000-00027. PMID 16052126